CLINICAL TRIAL: NCT03554304
Title: A Randomized, Double-Blind, Double-Dummy, Placebo- and Positive-Controlled, Crossover Study to Evaluate the Effect of WCK 5222 on the QT/QTc Interval in Healthy Volunteers
Brief Title: Evaluate the Effect of WCK 5222 on the QT/QTc Interval in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: W-5222-103
Record Dates: First submitted 2018-05-16; First posted 2018-06-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-05

CONDITIONS: QT/QTc Interval in Healthy Volunteers
MeSH Terms: interventions — cefepime-zidebactam; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- WCK 5222 (Experimental): WCK 5222 IV solution administered as either a 30- or 60-minute IV infusion)
  Interventions: Drug: WCK 5222; Drug: IV placebo matched to WCK 5222 / Moxifloxacin IV solution
- Placebo (IV placebo matched toWCK 5222IV solution) (Placebo Comparator): placebo capsule matched to moxifloxacin overencapsulated tablet IV placebo matched to WCK 5222 IV solution
  Interventions: Drug: IV placebo matched to WCK 5222 / Moxifloxacin IV solution
- Moxifloxacin 400-mg (Active Comparator): positive control
  Interventions: Drug: IV placebo matched to WCK 5222 / Moxifloxacin IV solution; Drug: Moxifloxacin 400-mg

INTERVENTIONS:
Drug: WCK 5222 — FEP-ZID IV solution administered as either a 30- or 60-minute IV infusion)
  Arms: WCK 5222
Drug: IV placebo matched to WCK 5222 / Moxifloxacin IV solution — Placebo (IV placebo matched to FEP-ZID IV solution) and
  1 placebo capsule matched to moxifloxacin overencapsulated tablet
  Other Names: Placebo capsule matched to moxifloxacin
Drug: Moxifloxacin 400-mg — Moxifloxacin 400-mg positive control (overencapsulated tablet)
  Arms: Moxifloxacin 400-mg

SUMMARY:
A Randomized, Double-Blind, Double-Dummy, Placebo- and Positive-Controlled, Crossover Study to Evaluate the Effect of WCK 5222 on the QT/QTc Interval in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index ≥18 to ≤33 kg/m2, inclusive.
2. Stable health based on a medical history without any major pathology/surgery in the 6 months

Exclusion Criteria:

1. An uninterpretable or abnormal screening electrocardiogram (ECG) indicating a second- or third-degree atrioventricular block
2. History of risk factors for torsades de pointes, including unexplained syncope, known long QT syndrome, heart failure, myocardial infarction, angina, or clinically significant abnormal laboratory assessments including hypokalemia, hypocalcemia, or hypomagnesemia.
3. A sustained supine systolic blood pressure >150 mm Hg or <90 mm Hg or a supine diastolic blood pressure >95 mm Hg or <50 mm Hg at Screening or Check-in (Day -1).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-10-06 (Actual)

PRIMARY OUTCOMES:
Incidence of delay in cardiac repolarization induced by WCK 5222 | 0-4 days
  as shown by analysis of the QT interval.

SECONDARY OUTCOMES:
Incidence of adverse events to assess tolerability at the supratherapeutic dose to be used in the thorough QT evaluation | 0-4 days
  Tolerability will be assessed by review of number of AEs
Incidence of AEs to assess the safety of high doses of single-dose administration of FEP-ZID | 0-4 days
  Safety will be assessed by review of adverse events (AEs), ECGs, and clinical laboratory safety test results

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No